CLINICAL TRIAL: NCT01807780
Title: Safety, Immunogenicity And Efficacy Of Vaccination In Military Personnel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Raffaele D'Amelio, Full Professor, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 01/2011 UGSAN
Record Dates: First submitted 2012-12-13; First posted 2013-03-08 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Vaccination Adverse Events; Vaccination Failure; Specific Antibody Response
MeSH Terms: interventions — Biological Monitoring

ARMS (1):
- single arm :vaccinated (Other): military personnel vaccinated with multiple vaccines and monitored about safety, immunogenicity and efficacy
  Interventions: Biological: biological monitoring

INTERVENTIONS:
Biological: biological monitoring

SUMMARY:
The purpose of this study is to determine if multiple vaccination in military personnel may be correlated with the appearance of poorly defined diseases as symptomatic multisyndrome, autoimmune or lymphoproliferative disorders. At the same time, considering possible interference between different vaccines, proteins and polysaccharides, living and inactivated, the study aims to assess the immunogenicity and efficacy also in relation to the specific Human Leucocyte Antigens (HLA) genetic structure.

ELIGIBILITY:
Inclusion Criteria:

* Military volunteers
* No recently immunized

Exclusion Criteria:

* Pregnancy
* Documented immunodepression
* Documented allergy or hypersensitivity to vaccines

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 262 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
immunomediated disorders related to multiple vaccination | three years

SECONDARY OUTCOMES:
efficacy of multiple vaccination | Three years
immunogenicity of multiple vaccination | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele D'Amelio, MD, Study Chair — sapienza università di roma
Locations (1):
- University of Roma La Sapienza, Roma, Italia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferlito C, Biselli R, Mariotti S, von Hunolstein C, Teloni R, Ralli L, Pinto A, Pisani G, Tirelli V, Biondo MI, Salerno G, Andreasi Bassi L, Lulli P, Autore A, Scagliusi A, Tomao E, Germano V, Picchianti Diamanti A, Caporuscio S, Milanetti F, Salemi S, Nisini R, D'Amelio R. Tetanus-diphtheria vaccination in adults: the long-term persistence of antibodies is not dependent on polyclonal B-cell activation and the defective response to diphtheria toxoid re-vaccination is associated to HLADRB1 *01. Vaccine. 2018 Oct 29;36(45):6718-6725. doi: 10.1016/j.vaccine.2018.09.041. Epub 2018 Sep 27. PMID 30269918